CLINICAL TRIAL: NCT00944645
Title: An Open Label, Randomized, 2-Period, Crossover Study to Establish the Definitive Bioequivalence of Niacin and MK0524 of 2 Sources of MK0524A Tablets
Brief Title: MK0524A Bioequivalence Study (0524A-059)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0524A-059; MK0524A-059; 2009_613
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin; MK-0524

ARMS (2):
- A (Active Comparator): MK0524A Source 1 (Phase III manufacturing site)
  Interventions: Drug: niacin (+) laropiprant (Source 1)
- B (Active Comparator): MK0524A Source 2 (commercial manufacturing site)
  Interventions: Drug: Comparator: niacin (+) laropiprant (Source 2)

INTERVENTIONS:
Drug: niacin (+) laropiprant (Source 1) — Single dose of MK0524A (ER Niacin/laropiprant 1000/20 mg) from Source 1 in one of two treatment periods.
  Arms: A
Drug: Comparator: niacin (+) laropiprant (Source 2) — Single dose of MK0524A (ER Niacin/laropiprant 1000/20 mg) from Source 2 in one of two treatment periods.
  Arms: B

SUMMARY:
This study will evaluate the definitive bioequivalence of tablets of MK0524A (1000 mg Extended Release (ER) Niacin/ 20 mg laropiprant) from two sources.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is willing to follow all study guidelines

Exclusion Criteria:

* Subject has or has a history of any disease or condition that might confound the results of the study or make participation unsafe

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK0524A Phase III Tablet Then MK0524A New Site Tablet: MK0524A Phase III tablet: MK0524A (1000 mg ER Niacin/20 mg MK0524) Phase III tablet (Source 1)/MK0524A New Site tablet: MK0524A (1000 mg ER Niacin/20 mg MK0524) tablet from new manufacturing site (Source 2)
- MK0524A New Site Tablet Then MK0524A Phase III Tablet: MK0524A New Site tablet: MK0524A (1000 mg ER Niacin/20 mg MK0524) tablet from new manufacturing site (Source 2)/ MK0524A Phase III tablet: MK0524A (1000 mg ER Niacin/20 mg MK0524) Phase III tablet (Source 1)
Period: Period 1
Arm/Group | MK0524A Phase III Tablet Then MK0524A New Site Tablet | MK0524A New Site Tablet Then MK0524A Phase III Tablet
Started | 94 | 94
Completed | 94 | 94
Not Completed | 0 | 0
Period: Period 2
Arm/Group | MK0524A Phase III Tablet Then MK0524A New Site Tablet | MK0524A New Site Tablet Then MK0524A Phase III Tablet
Started | 94 | 94
Completed | 86 | 85
Not Completed | 8 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes all participants from Both treatment groups; MK0524A Phase III tablet and MK0524A New Site tablet
Arm/Group | All Participants
Number analyzed (Participants) | 188
Age, Continuous [Mean (Full Range); unit: years] | 38.5 (1) [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 96
Height [Mean (Full Range); unit: Centimeters] | 166.6 [140 to 190]
Weight [Mean (Full Range); unit: Kilograms] | 71.6 [48.4 to 101]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Nicotinuric Acid
Description: Measure of rate of absorption of ER niacin
Time Frame: Predose and up to 24 hours postdose
Population: The Hodges-Lehmann estimator was used to analyze nicotinuric acid Cmax and uses only subjects with data available on both treatment periods. 188 subjects were randomized,17 subjects discontinued, 26 subjects were inadvertently overdosed with 5 tablets of MK0524A 1000 mg/20 mg, reducing the available subject population for analysis to 145.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- MK0524A New Site Tablet: MK0524A (1000 mg ER Niacin/20 mg laropiprant) tablet from new manufacturing site (Source 2)
- MK0524A Phase III Tablet: MK0524A (1000 mg ER Niacin/20 mg laropiprant) Phase III tablet (Source 1)
Arm/Group | MK0524A New Site Tablet | MK0524A Phase III Tablet
Number analyzed (Participants) | 145 | 145
ng/mL | 1190 [956 to 1610] | 1260 [948 to 1660]
Statistical Analysis 1: Comparison: MK0524A New Site Tablet vs MK0524A Phase III Tablet; MK0524A (1000 mg ER Niacin/20 mg MK-laropiprant) tablet from new manufacturing site (Source 2) MK0524A (1000 mg ER Niacin/20 mg MK-laropiprant) Phase III tablet (Source 1); Test type: Non-Inferiority or Equivalence — Primary research hypothesis I: The Cmax of nicotinuric acid (NUA) following the administration of MK0524A (ER niacin 1000 mg/ laropiprant 20 mg) tablets from 2 manufacturing sites is similar (i.e., the true GMR of NUA Cmax is contained within the bioequivalence interval (0.80, 1.25)); Geometric Mean Ratio = 0.98, 90% CI [0.93 to 1.03]

2. Primary Outcome: Total Amount of Urinary Excretion of Niacin and Its Metabolites
Description: Measure of extent of absorption of ER niacin
Time Frame: Predose and up to 96 hours postdose
Population: A linear mixed effect model was used to analyze total amount of urinary excretion of niacin and its metabolite and uses data available from at least one treatment period. 157 subjects had data from the treatment of MK0524A New Site Tablet, and 161 subjects had data from the treatment of MK0524A Phase III Tablet
Measure: Median (Standard Deviation); unit: micro mole
Arm/Group | MK0524A New Site Tablet | MK0524A Phase III Tablet
Number analyzed (Participants) | 157 | 161
micro mole | 5280 (1894) | 5470 (1330)
Statistical Analysis 1: Comparison: MK0524A New Site Tablet vs MK0524A Phase III Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Primary research hypothesis II: The total urinary excretion of niacin and niacin metabolites following the administration of MK0524 (ER niacin 1000 mg/ laropiprant 20 mg) tablets from 2 manufacturing sites is similar (i.e., the true GMR of total urinary excretion of niacin and its metabolites is contained within the bioequivalence interval (0.80, 1.25)); Geometric Mean Ratio = 0.94, 90% CI [0.89 to 0.98]

3. Primary Outcome: Area Under Curve (AUC 0-infinity) of Laropiprant
Description: Measure of extent of absorption of laropiprant
Time Frame: Predose and up to 48 hours postdose
Population: A linear mixed effect model was used to analyze laropiprant AUC0-infinity and uses data available from at least one treatment period. 166 subjects had data from the treatment of MK0524A New Site Tablet, and 167 subjects had data from the treatment of MK0524A Phase III Tablet
Measure: Median (Standard Deviation); unit: Micro Molar times Hour
Arm/Group | MK0524A New Site Tablet | MK0524A Phase III Tablet
Number analyzed (Participants) | 166 | 167
Micro Molar times Hour | 6.36 (3.01) | 6.37 (2.66)
Statistical Analysis 1: Comparison: MK0524A New Site Tablet vs MK0524A Phase III Tablet; Group B: MK0524A (1000 mg ER Niacin/20 mg MK-laropiprant) tablet from new manufacturing site (Source 2) Group A: MK0524A (1000 mg ER Niacin/20 mg MK-laropiprant) Phase III tablet (Source 1); Test type: Non-Inferiority or Equivalence — Primary research hypothesis III: The AUC0-infinity of laropiprant following the administration of MK0524A (ER niacin 1000 mg/ laropiprant 20 mg) tablets from 2 manufacturing sites is similar (i.e., the true GMR of MK0524 AUC0-∞ is contained within the bioequivalence interval (0.80, 1.25)); Geometric Mean Ratio = 1.00, 95% CI [0.95 to 1.05]

4. Primary Outcome: Maximum Concentration (Cmax) of Laropiprant
Description: Measure of rate of absorption of laropiprant
Time Frame: Predose and up to 48 hours postdose
Population: A linear mixed effect model was used to analyze laropiprant Cmax and uses data available from at least one treatment period. 166 subjects had data from the treatment of MK0524A New Site Tablet, and 167 subjects had data from the treatment of MK0524A Phase III Tablet.
Measure: Median (Standard Deviation); unit: micro Molar
Arm/Group | MK0524A New Site Tablet | MK0524A Phase III Tablet
Number analyzed (Participants) | 166 | 167
micro Molar | 0.988 (0.563) | 0.975 (0.466)
Statistical Analysis 1: Comparison: MK0524A New Site Tablet vs MK0524A Phase III Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Primary research hypothesis IV: The Cmax of laropiprant following the administration of MK0524A (ER niacin 1000 mg/ laropiprant 20 mg) tablets from 2 manufacturing sites is similar (i.e., the true GMR of MK0524 Cmax is contained within the bioequivalence interval (0.80, 1.25)); Geometric Mean Ratio = 1.02, 95% CI [0.96 to 1.09]

ADVERSE EVENTS:
Arm/Group | MK0524A Phase III Tablet | MK0524A New Site Tablet
Serious Adverse Events (participants affected / at risk) | 0/188 | 2/188
Other Adverse Events (participants affected / at risk) | 98/188 | 100/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0524A Phase III Tablet (N=188) | MK0524A New Site Tablet (N=188)
Hematemesis (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0524A Phase III Tablet (N=188) | MK0524A New Site Tablet (N=188)
Palpitations (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 2 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1
Eye Irritation (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Defaecation Urgency (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 2
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 13 | 11
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 6
Chest Discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Influenza Like Illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Herpes Simplex (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Viral Infection (Infections and infestations) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 12 | 14
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Amylase Increased (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Helicobacter Pylori Identification Test Positive (Investigations) | 1 | 0
Lipase Increased (Investigations) | 0 | 1
Occult Blood Positive (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 10 | 7
Headache (Nervous system disorders) | 15 | 20
Paraesthesia (Nervous system disorders) | 16 | 16
Syncope (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Bladder Pain (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 19
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 69 | 70
Vasodilatation (Vascular disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.